CLINICAL TRIAL: NCT04307628
Title: Response of Gut Microbiota and Cardiometabolic Biomarkers to Consumption of Walnuts
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study logistics still being worked out. On hold for now.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1562149
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Healthy; Normal Weight; Overweight; Obese
MeSH Terms: conditions — Overweight; Obesity | interventions — PR-10 protein, walnut birch pollen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walnut (Active Comparator): Eat 2 ounces of walnuts provided by the study. Eating any other nuts is to be avoided. Background diet will be low in polyphenols.
  Interventions: Other: Walnut
- Nut-Free (Placebo Comparator): Eating any other nuts is to be avoided. Background diet will be low in polyphenols.
  Interventions: Other: Nut-Free

INTERVENTIONS:
Other: Walnut — Study participants will eat 2 ounces of walnuts each day.
  Arms: Walnut
Other: Nut-Free — Study participants will not eat nuts.
  Arms: Nut-Free

SUMMARY:
The researchers will investigate blood and fecal responses in qualified study participants after eating walnuts for 4 weeks compared to not eating walnuts for 4 weeks. The two dietary interventions will be separated by a 4 week washout period. The order of diets will be random; study participants will complete both interventions. Dietary modifications will be part of the study protocol.

DETAILED DESCRIPTION:
The researchers hypothesize that walnut consumption will induce changes in fecal metagenome, identifiable walnut-derived bioactives (urolithins) and other microbial-derived products (short-chain fatty acids and secondary bile acids). The researchers hypothesize that walnut consumption will result in improvements to blood lipid profiles, including decreased total and LDL-cholesterol; increased HDL-related cholesterol efflux capacity and antioxidant protection; and decreased inflammatory biomarkers relative to control diet. The researchers hypothesize changes in cardiometabolic health biomarkers will be correlated with food bioactive metabolites and/or fecal metagenome. Pathway analysis will identify metabolic pathways differentially regulated by walnut-derived bioactives and walnut-responsive microbial genes.

ELIGIBILITY:
Inclusion Criteria:

Generally healthy men and women between 20-65 years of age and BMI range of 20.0-34.9 kg/m2 will be recruited from the Davis - Sacramento metropolitan area. Enrolled subjects must be willing to consume 2 ounces (approximately 1/2 cup) of walnuts daily and modify their diet to avoid eating walnuts and other nuts, and foods or beverages high in polyphenols (a list will be provided) during study enrollment . Adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant or lactating women, women planning to become pregnant in the next four months and prisoners will be specifically excluded. Screening will take place by phone interview and through in-person screening and consent, including anthropometric and biochemical assessments and health history questionnaires.

Exclusion Criteria:

* Allergy to walnuts or other nuts
* Eating more than 25 grams of fiber per day, assessed by the Block Dietary-Fruit-Vegetable-Fiber Screener©
* Taking medications or supplements known to affect metabolism or gut microbiota composition (i.e. Metformin, statins, antibiotics within the past 3 months, fiber supplements, probiotics, and others)
* Documented chronic diseases including diabetes, renal or liver disease, metabolic syndrome, active cancer, MI or stroke, history of gastric bypass or GI disease (e.g. Crohn's Disease, Irritable Bowel Disease, diverticulosis/diverticulitis,etc)
* Smoker or living with a smoker, including vaporizer and/or electronic cigarettes.
* Illicit drug use, cannabis usage, or consuming >1 alcoholic drink/day
* Extreme dietary or exercise patterns; vegan diet.
* Recent weight fluctuations (>10% in the last 6 months)
* Taking prescription lipid medications or supplements that may affect lipoprotein metabolism (i.e. >1 g of fish oil/day, antioxidant supplements)
* Taking exogenous hormones (e.g. hormonal birth control)
* Poor venous access
* Unwillingness to comply with study protocols

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Assessing the influence of walnuts on the fecal metagenome | Through study completion, an average of 12 weeks
  Changes in fecal metagenomics will be assessed via Illumina sequencing
Assessing the influence of walnuts on fecal secondary bile acids | Through study completion, an average of 12 weeks
  Fecal secondary bile acids will be measured by LC-QTOF/MS
Assessing the influence of walnuts on fecal short-chain fatty acids | Through study completion, an average of 12 weeks
  Short-chain fatty acids in fecal matter will be measured by LC-MS/MS
Urolithins measured in plasma by UPLC/MS | Through study completion, an average of 12 weeks
  Measure for changes in the levels of urolithins in separated plasma; measured in units of ug/uL. Blood will be assessed at each of the 4 study visits.
Fecal calprotectin will be measured by ELISA | Through study completion, an average of 12 weeks
  Measure for changes in the levels of calprotectin in collected fecal matter; measured in units of ug/g. Feces will be assessed at each of the 4 study visits.

SECONDARY OUTCOMES:
Assessing the influence of walnuts on blood lipid measurements | Through study completion, an average of 12 weeks
  Measure for changes in the levels of HDL and LDL in separated plasma; measured in units of mg/dL. Blood will be assessed at each of the 4 study visits
Assessing the influence of walnuts on paraoxonase-1 (PON-1) activity | Through study completion, an average of 12 weeks
  Measure for changes in PON-1 activity in separated plasma at each study of the 4 study visits. Activity will be calculated based on linear rates of hydrolysis of phenyl acetate to phenol
Assessing the influence of walnuts on cholesterol ester transfer protein activity (CETP) | Through study completion, an average of 12 weeks
  Changes in CETP activity will be measured at each of the 4 study visits. The isolated plasma will be co-incubated with donor and acceptor molecules using a commercially available assay kit.
Assessing the influence of walnuts on hsCRP will be measured in blood | Through study completion, an average of 12 weeks
  hsCRP will be measured in blood at each study visit
Assessing the influence of walnuts on SAA will be measured in blood | Through study completion, an average of 12 weeks
  SAA will be measured in blood at each study visit
Assessing the influence of walnuts on circulating cytokines | Through study completion, an average of 12 weeks
  ICAM and VCAM will be measured in blood at each study visit using a commercially available ELISA kit.
Assessing the influence of walnuts on peripheral blood mononuclear cells (PBMC) using ex vivo stimulation assays | Through study completion, an average of 12 weeks
  In-vitro: media from LPS stimulated monocytes will be used to measure gene expression and cytokines Measurement of changes in PBMC derived cytokines as a marker of inflammation at each of the 4 study visits. Assessment will be based on an increase or decrease in concentration in pg/ml.
Dietary record analysis | Through study completion, an average of 12 weeks
  Use a computer program to check for study dietary requirements. Subjects are to avoid olives and olive containing products during study protocol periods. This will be done using a subject self-recorded 3-day food record submitted to study personnel.
Anthropometric measurements | Through study completion, an average of 12 weeks
  Measure waist (cm) and hip circumference (cm) before the start of drawing blood on study day protocols.
Measure for changes in weight | Through study completion, an average of 12 weeks
  Measure weight (kg) before the start of drawing blood on study day protocols
Measure for changes in blood pressure | Through study completion, an average of 12 weeks
  Measure blood pressure (mmHg) before the start of drawing blood on study day protocols

CONTACTS AND LOCATIONS:
Overall Officials: Francene M Steinberg, PhD, RD, Principal Investigator — University of California, Davis
Locations (1):
- Ragle Human Nutrition Research Center, Davis, California, United States